CLINICAL TRIAL: NCT05032846
Title: Intra-operative Ultrasound Guided Laparoscopic Ovarian Cystectomy (UGLOC) as a Method of Fertility Preservation in the Management of Benign Ovarian Cysts: Randomised Controlled Trial
Brief Title: Intra-operative Ultrasound Guided Laparoscopic Ovarian Cystectomy as a Method of Fertility Preservation
Acronym: UGLOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 290747
Record Dates: First submitted 2021-08-16; First posted 2021-09-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Benign Ovarian Cyst
Keywords: Intraoperative ultrasound; Fertility Preservation; Benign Ovarian Cyst; Anti-Mullerian Hormone

STUDY DESIGN:
Intervention Model Description: Non-blinded randomised clinical trial
Masking Description: Non-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Laparoscopic Ovarian Cystectomy (Experimental): During surgical resection of the ovarian cyst, a clinician with experience of ultrasound and laparoscopy will perform an ultrasound scan during surgery to resect cyst tissue only and preserve healthy ovarian tissue.
  Interventions: Procedure: Ultrasound guided laparoscopic ovarian cystectomy
- Laparoscopic Ovarian Cystectomy (Active Comparator): A laparoscopic ovarian cystectomy will be performed without ultrasound guidance. This is currently standard clinical practice.
  Interventions: Other: Laparoscopic Ovarian Cystectomy

INTERVENTIONS:
Procedure: Ultrasound guided laparoscopic ovarian cystectomy — Laparoscopic ovarian cystectomy to be performed under intra-operative ultrasound guidance.
  Arms: Ultrasound Guided Laparoscopic Ovarian Cystectomy
Other: Laparoscopic Ovarian Cystectomy — Laparoscopic Ovarian Cystectomy will be performed as standard clinical practice.
  Arms: Laparoscopic Ovarian Cystectomy

SUMMARY:
Title:

Intra-operative ultrasound guided laparoscopic ovarian cystectomy (UGLOC) as a method of fertility preservation in the management of benign ovarian cysts.

Background:

Approximately 10% of women in the United Kingdom (UK) will undergo surgery for the presence of an ovarian mass during their lifetime. Ovarian surgery, however, is not without risks and can potentially harm healthy ovarian tissue surrounding the cyst, resulting in reduced reproductive potential (the ability of the ovary to produce eggs for fertilisation). Surgical methods to preserve healthy ovarian tissue and improve the chances of successful pregnancy post-operatively are known as Fertility Preserving Surgery (FPS). Evidence suggests that a novel approach of FPS involving the removal of an ovarian cyst performed under ultrasound guidance improves the differentiation between the healthy ovarian tissue and the ovarian cyst. As such, the surgeon can remove the cyst alone, whilst limiting disruption to the healthy surrounding ovarian tissue.

Aim:

The purpose of this study is to assess if surgical removal of an ovarian cyst performed under ultrasound guidance improves the reproductive potential of the ovaries, when compared to surgery performed without ultrasound guidance.

Eligibility

All patients of reproductive age (18-45 years old) with ultrasound features suggestive of a benign ovarian cyst requiring surgical treatment (removal of the cyst). Patients diagnosed with benign ovarian cysts, deemed to be non -harmful to the patient if left untreated, of the following classifications can be included in the study: dermoid, simple cyst, serous cystadenoma, mucinous cystadenoma or endometrioma.

Design:

A multicentre randomised controlled trial. Women across Imperial College London Healthcare and University College London Trusts will be allocated to a surgical treatment group at random: 1) laparoscopic ovarian cystectomy performed without ultrasound guidance (control group) or 2) ultrasound guided laparoscopic ovarian cystectomy performed with ultrasound guidance (fertility preservation surgery: intervention group).

Duration:

3 years

DETAILED DESCRIPTION:
Background:

The use of intra-operative ultrasound has been widely implemented amongst other specialties. However, within gynaecological surgery, it is not as commonly recognized, despite evidence that it can be used as an adjunct to improving minimally invasive surgical techniques. This is primarily due to the improved visualization of the operative field, which can assist more technically difficult surgical procedures, thus minimizing intra-operative complications. The application of ultrasound guidance within gynaecological procedures have included predominantly ovarian cyst aspiration, in vitro fertilization and removal or insertion of intra-uterine devices. Although pre-operative imaging provides procedural planning, it cannot compare to the information gained from real time imaging. For example, in previous studies, intra-operative ultrasound detected more myomas during myomectomy than pre-operative transvaginal imaging. Furthermore, it provides the potential to assess lesion margins, ensuring resection of pathology is complete with negligible damage to surrounding healthy tissues. This is consistent with a recent systematic review, which also demonstrated that albeit a novel technique, amongst various case series, pathology can be safely resected without incurring injury to healthy reproductive tissue. Therefore, intra-operative ultrasound has the potential to improve surgical accuracy, reduce complications and improve patient safety. The application of intra-operative ultrasound as an adjunct to fertility sparing surgery has not been widely researched, with only a few case series reporting surgical outcomes on patients undergoing treatment for pre-malignant or malignant pathology. The aim of this study therefore, is to determine the efficacy of this surgical technique in the management of benign pathology, including the surgical resection of ovarian cysts.

Hypothesis:

Intra-operative ultrasound will prove a significant method of fertility preservation surgery, as measured by a significantly reduced decrease in Anti-Mullerian Hormone (AMH) and antral follicle count (AFC) at 3 and 6 months post-operatively, when compared to the control group.

Study Design:

This will be a multi-centre prospective cohort study carried out as a non-blinded randomised controlled trial. Women will be allocated to either a control group of laparoscopic ovarian cystectomy performed without ultrasound guidance, or to the experimental ultrasound guided laparoscopic ovarian cystectomy (UGLOC) group. All surgeons operating and women recruited to the study will be aware of which group they have been allocated to from the beginning of their participation to the study. The research team aims for equal sample sizes in both groups.

Recruitment:

Women referred to the outpatient gynaecology clinic with a suspected ovarian cyst will be asked about their clinical history and undergo a pelvic transvaginal ultrasound scan (2D and 3D ultrasonography) as part of routine clinical care. If an ovarian cyst is seen on ultrasound, it will be assessed according to local protocols based on simple descriptors and International Ovarian Tumour Analysis (IOTA) simple rules. Depending on the severity of symptoms, nature of the cyst and fulfilment of the inclusion criteria and if the woman is suitable for surgical management, she will then be invited to participate in the study. Participants will be recruited from various general gynaecology clinics, as well as specialist clinics including: ovarian cyst clinic, the IOTA and Rapid access clinics across Imperial and University College London Hospital.

Following consent of participation, the woman will be assigned to either a control or experimental group. A separate research group, not directly affiliated with the project will perform the randomisation process. The research group will print x "control group" labels and x "experimental group," in which each label is then sealed into an individual envelope. All envelopes will be numbered and issued in sequence. During the recruitment process, once the participant has given consent to participate in the trial, a member of the research team will select the envelope in sequence, which will then assign the participant to a group. This will prevent the person performing the randomisation from selecting another envelope if they are not happy with the group allocation.

For this study, it will not be necessary to postpone diagnostic procedures or treatment, and participation will not influence normal treatment.

Surgical Intervention:

The same surgeons will operate on women in both the control and experimental group. This will aim to exclude bias which may otherwise attribute findings to the surgeon operating. Surgery will be performed at Imperial Healthcare NHS Trusts and at the University College London Hospitals NHS Foundation Trust by an experienced clinician.

Data Collection:

The research team will collect the following data: Participant demographics including age, BMI, gravida, parity and gynaecological surgical history. Pre-operative data will include findings from the diagnostic transvaginal scan and measure of ovarian reserve: AMH and AFC. Intra-operative data will include transvaginal findings during surgery (in the experimental group only), such as cyst location and size or any new lesions noted. Residual ovarian volume post cystectomy will also be measured intraoperatively. Histology data will include the histological diagnosis of the ovarian cyst and volume of normal ovarian tissue excised during the cystectomy measured as per margins in mm. Outcomes following surgery including duration of surgery (mins), length of hospital stay (days) and post operative complications will be recorded.

Follow up:

Post-operatively, participants will return to their respective hospital gynaecology clinic responsible for the care and management of the ovarian cyst for follow up at 3 and 6 months. During the appointment a blood test will be taken to assess ovarian reserve by measuring the AMH level. The outpatient gynaecology nurse in clinic or research staff will be responsible for taking the blood sample and will only require one EDTA bottle (yellow top) to be filled (20-40mls). The blood samples will be processed by Imperial College Healthcare Trust laboratories or University College London Hospitals NHS Foundation Trust, depending on the site taken, and will be discarded as per local protocol once the AMH has been determined. There are no specific storage or transfer requirements outside of normal practice. Therefore, samples will be 'podded' to the labs once taken in the usual way. In addition, an ultrasound will be performed during the follow up appointment by an experienced gynaecology specialist trainee or Consultant to assess the AFC and preserved ovarian volume of tissue remaining. Any incidental findings identified on ultrasound scan of gynaecological pathology, will be managed by the responsible clinician and the participants GP will be informed by letter. Follow up appointments should take approximately 20 minutes. The two blood tests and two ultrasound scans carried out during the follow up process are considered standard clinical practice, and therefore not considered additional investigations for the purpose of this research study.

The majority of participants are likely to be discharged following their 2nd clinic appointment 6 months post- surgery, whereby no further involvement in the study is required. If a participant becomes pregnant during the follow up period, clinic appointments will be deferred to 3 and 6 months post-partum.

ELIGIBILITY:
Inclusion Criteria:

All patients of reproductive age with a diagnosis of a benign ovarian cyst requiring surgical management.

This includes cysts defined as dermoid, teratoma, simple cyst, functional, serous cystadenoma or mucinous cystadenoma from the initial diagnostic ultrasound.

A strict criterion for the US diagnostic features will include the following:

* Cyst size ≥3cm; ≤10cm
* The International Ovarian Tumour Analysis for benign features (IOTA B) only:

  * Unilocular
  * Solid components: largest diameter ≤7mm
  * Acoustic shadows
  * No blood flow
  * Smooth multilocular cyst: largest diameter ≤10cm

Specifically:

* Pregnant patients can be included but will be analysed separately
* For patients selected for surgery, delay of surgery is not an exclusion criterion for this study, but for selected objectives we will use only those patients in whom surgery was performed within 180 days after the ultrasound examination
* With regards to age, patients can be selected only if 18-50 years old.
* Patients whom only underwent transabdominal scanning can be included in the study, but will be analysed separately

Exclusion Criteria:

* Cysts that are deemed to be clearly physiological and less than <3 cm in maximum diameter are not eligible for inclusion
* Cysts ≥11cm in maximum diameter
* Non-adnexal masses e.g. peritoneal inclusion cysts (where diagnosis is certain).
* Any cyst with features of malignancy
* The denial or withdrawal of written informed consent
* Women of post- menopausal or peri-menopausal status

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone (AMH) (pmol/L) | 3 years
  Post operative AMH level will be measured at 3 and 6 months post surgery.
Antral Follicle Count (AFC) (n) | 3 years
  Post operative AFC will be measured at 3 and 6 months post surgery.

SECONDARY OUTCOMES:
Length of hospital stay (days) | 3 years
  Surgical outcomes will be determined such as the length of hospital stay measured in days in the control and experimental group.
Presence of intra-operative cyst rupture (Yes/No) | 3 years
  During the procedure, it will be determined whether or not there has been a cyst rupture, whereby cyst contents have dispersed into the abdominal cavity in the control and experimental group.
Duration of surgery (minutes) | 3 years
  The duration of surgery will be measured in the control and experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Yazbek, MD, Principal Investigator — Imperial College London Healthcare Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It will not be necessary to share individual participant data (IPD) with other researchers outside of the immediate research team. The only members with access to the information will be the PI (Joseph Yazbek) and the tudy Co-ordinator (Lorraine Kasaven).

REFERENCES:
- [Derived] Kasaven LS, Jones BP, Ghaem-Maghami S, Verbakel JYJ, El-Bahrawy M, Saso S, Yazbek J. Study protocol for a randomised controlled trial on the use of intraoperative ultrasound-guided laparoscopic ovarian cystectomy (UGLOC) as a method of fertility preservation in the management of benign ovarian cysts. BMJ Open. 2022 Jul 14;12(7):e060409. doi: 10.1136/bmjopen-2021-060409. PMID 35835531

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT05032846/SAP_000.pdf
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05032846/ICF_001.pdf